CLINICAL TRIAL: NCT04068987
Title: Parametric Mapping in Paediatric Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Kenneth CHEUNG, Associate Consultant, Hong Kong Children's Hospital
Other Study IDs: HKCH-REC-2019-014
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Disease; Pediatric Disease; Cardiomyopathies; Congenital Disorders
Keywords: magnetic resonance imaging; parametric mapping
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers
  1. Recruited from the public
  2. Patients who have scheduled imaging scans for non-cardiac reasons and without a prior history or suspected history of cardiac disease
  Interventions: Diagnostic Test: MRI parametric mapping
- Children undergoing clinically indicated cardiac MRI: Patients who are scheduled to have a clinically indicated cardiac MRI
  Interventions: Diagnostic Test: MRI parametric mapping

INTERVENTIONS:
Diagnostic Test: MRI parametric mapping — Magnetic resonance (MR) sequences (T1 mapping, T2 mapping, T2* mapping, ECV mapping) to determine the MR signal characteristics of the body

SUMMARY:
Magnetic resonance imaging (MRI) is increasingly an important tool for diagnosis and management of cardiac diseases in children.

One of the uses of MRI is tissue characterisation, in which the signal characteristics of the cardiac muscle (myocardium) can be determined with special techniques, known as parametric mapping.

There is increasing evidence that parametric mapping may be able to identify regions of scarring in the myocardium, or detection of oedema/inflammation in the setting. This in turn can help predict disease course and add value to the management of patients.

There is also evidence that other structures that are visualised in parametric mapping aside from the heart (e.g. liver and spleen) can also help improve diagnostic accuracy and guide management.

Currently the majority of studies describing the use of parametric mapping is focused on adults, with limited data on its use in children.

The parametric mapping values can also differ amongst different machines, so calibration with normal subjects are also required.

DETAILED DESCRIPTION:
Magnetic resonance Imaging (MRI) can provide tissue characterisation without radiation and need for invasive biopsy.

Parametric mapping techniques (T1 mapping, extracellular volume fraction, T2 mapping, T2* mapping) are methods of quantitative analysis of tissue properties, and are currently commercially available.

T1 mapping, extracellular volume fraction (ECV) and T2* mapping provides knowledge about the tissue properties of the myocardium, interstitium and adjacent structures,and can provide information for diagnosis of fibrosis, inflammatory and infiltrative diseases.

T2 mapping is useful for assessing oedema, which may be useful in monitoring disease activity such as myocarditis.

Parametric mapping has proven clinical utility in iron deposition, amyloid disease, Anderson-Fabry disease and myocarditis.

In addition to assessment of cardiac muscle, tissue characterisation can also be performed in adjacent organs that are included in the field of view of parametric mapping (e.g. liver and spleen).

Parametric mapping may provide important diagnostic information for decision making, patient monitoring and management planning.

The investigators aim to

1. recruit healthy volunteers as controls to establish normal local reference ranges for parametric mapping values
2. recruit patients undergoing clinically indicated cardiac MRI to perform parametric mapping, and compare the parametric mapping values between normal controls and patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Paediatric patients <=18 years of age with suspected or confirmed cardiac disease undergoing clinically indicated MRI

Exclusion Criteria:

* Unstable or uncooperative patients that cannot tolerate MRI
* Patients with contraindications for MRI (e.g. patients with implanted devices that are not MRI compatible)

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Healthy Volunteers
  2. Patients with suspected or confirmed cardiac disease undergoing clinically indicated MRI.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Parametric mapping values of normal subjects and patients | through study completion, up to 2 years
  Parametric mapping values are generated upon completion of the MR sequence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Anonymised patient data can be shared upon request

REFERENCES:
- [Background] Messroghli DR, Moon JC, Ferreira VM, Grosse-Wortmann L, He T, Kellman P, Mascherbauer J, Nezafat R, Salerno M, Schelbert EB, Taylor AJ, Thompson R, Ugander M, van Heeswijk RB, Friedrich MG. Clinical recommendations for cardiovascular magnetic resonance mapping of T1, T2, T2* and extracellular volume: A consensus statement by the Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI). J Cardiovasc Magn Reson. 2017 Oct 9;19(1):75. doi: 10.1186/s12968-017-0389-8. PMID 28992817
- [Background] Kim PK, Hong YJ, Im DJ, Suh YJ, Park CH, Kim JY, Chang S, Lee HJ, Hur J, Kim YJ, Choi BW. Myocardial T1 and T2 Mapping: Techniques and Clinical Applications. Korean J Radiol. 2017 Jan-Feb;18(1):113-131. doi: 10.3348/kjr.2017.18.1.113. Epub 2017 Jan 5. PMID 28096723
- [Background] Riesenkampff E, Messroghli DR, Redington AN, Grosse-Wortmann L. Myocardial T1 mapping in pediatric and congenital heart disease. Circ Cardiovasc Imaging. 2015 Feb;8(2):e002504. doi: 10.1161/CIRCIMAGING.114.002504. No abstract available. PMID 25657297
- [Background] Anderson LJ. Assessment of iron overload with T2* magnetic resonance imaging. Prog Cardiovasc Dis. 2011 Nov-Dec;54(3):287-94. doi: 10.1016/j.pcad.2011.07.004. PMID 22014495